CLINICAL TRIAL: NCT00522496
Title: Proteomics of Severe Traumatic Brain Injury: A Feasibility Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Collaborators: Canadian Intensive Care Foundation (Other)
Responsible Party: David Zygun Principal Investigator, University of Calgary
Other Study IDs: 20216
Record Dates: First submitted 2007-08-27; First posted 2007-08-29 (Estimated); Last update posted 2009-02-24 (Estimated); Status verified 2009-02

CONDITIONS: Brain Injuries, Traumatic
Keywords: Craniocerebral trauma; matrix metalloproteinase; microdialysis
MeSH Terms: conditions — Brain Injuries, Traumatic; Craniocerebral Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to:

1. Determine the temporal course of matrix metalloproteinase (MMP) expression in patients wiht severe traumatic brain injury
2. Determine the temporal course of the expression of MMP-related inflammatory mediators of secondary injury in patients with severe traumatic brain injury
3. Describe the association of physiological changes and standard microdialysis analyte measures (lactate, pyruvate, lactate/pyruvate ratio, and glucose) to MMP and neuroinflammatory marker concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years of age or older
* Patient has GCS less than 9
* Patient requires intracranial pressure monitoring
* Patient life expectancy greater than 72 hours

Exclusion Criteria:

* Patient's TBI is greater than 24 hours old
* Patient is less than 18 years of age
* Patient does not require intracranial pressure monitoring
* Patient has life expectancy less than 72 hours
* Patient has GCS greater or equal to 9
* Patient is currently enrolled in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients referred to Foothills Medical Centre, the regional trauma centre for Southern Alberta
Sampling Method: Non-Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2007-07; Study Completion 2009-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Zygun A David, MD, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada